CLINICAL TRIAL: NCT06893237
Title: The Effect of Virtual Reality Goggles and Distraction Cards Applied to Children Aged 6-12 Years During Inhaler Therapy on Physiological Parameters and Anxiety: a Randomised Controlled Study
Brief Title: The Effect of Virtual Reality Goggles and Distraction Cards Applied to Children Aged 6-12 Years During Inhaler Therapy on Physiological Parameters and Anxiety
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Tuğba Karakaya, Principal investigator, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UskudarU-SBE-TK-02
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Respiratory Infections, Acute; Respiratory Tract Diseases
Keywords: inhalation therapy; child; virtual reality glasses; anxiety; distraction of attention
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Tract Diseases; Anxiety Disorders | interventions — Respiratory Therapy

STUDY DESIGN:
Intervention Model Description: three groups with traditional therapy control group.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- virtual reality group (Experimental): Video recording will be started after the consent is obtained. Physical parameters (peak heart rate, respiratory rate, oxygen saturation) and anxiety of the child will be measured and recorded 1 minute before the procedure. Then, the child will be fitted with virtual reality goggles and inhalation treatment will be started by watching the aquarium and sea creatures video. Inhalation treatment will last for 10 minutes with the most appropriate air flow rate of 6-8 L/min. Then, the virtual reality goggles will be removed and the child's physiological parameters and anxiety will be measured and recorded again after 1 minute. For participants who want to participate in the study but do not approve the video recording, the evaluations will be made by a nurse independent of the study.
  Interventions: Other: virtual reality goggles and inhalation treatment
- group of distraction cards (Experimental): Video recording will be started after the consent is obtained. One minute before the procedure, the child's physical parameters (peak heart rate, respiratory rate, oxygen saturation) and anxiety will be measured and recorded. Then, the child will be shown the distraction cards and inhalation treatment will be started simultaneously. Playing with the distraction cards will continue for 10 minutes until the end of inhalation treatment. Then, the use of toys will be terminated and the child's physiological parameters and anxiety will be recorded after 1 minute. Video recording will be terminated. For participants who want to participate in the study but do not consent to be video recorded, the evaluations will be carried out by a nurse independent of the study.
  Interventions: Other: distraction cards and inhalation therapy
- control group (Active Comparator): Video recording will be started after the consent is obtained. Physical parameters (peak heart rate, respiratory rate, oxygen saturation) and anxiety of the child will be measured and recorded 1 minute before the procedure. Then, inhalation treatment will be started with routine service practice. The child will receive inhalation treatment for 10 minutes. Physiological parameters and anxiety will be measured and recorded again 1 minute after the procedure. Video recording will be terminated. For participants who want to participate in the study but do not approve the video recording, the evaluations will be made by a nurse independent of the study.
  Interventions: Other: inhalation therapy

INTERVENTIONS:
Other: virtual reality goggles and inhalation treatment — Video recording will be started after the consent is obtained. One minute before the procedure, the child's physical parameters (peak heart rate, respiratory rate, oxygen saturation) and anxiety will be measured and recorded. Then, the child will be fitted with virtual reality goggles and inhalation treatment will be started by watching the aquarium and sea creatures video. Inhalation treatment will last for 10 minutes with the most appropriate air flow rate of 6-8 L/min. Then, the virtual reality goggles will be removed and the child's physiological parameters and anxiety will be measured and recorded again after 1 minute. For participants who want to participate in the study but do not approve the video recording, the evaluations will be made by a nurse independent of the study.
  Arms: virtual reality group
Other: distraction cards and inhalation therapy — After the consent is obtained, the video recording will be started. 1 minute before the procedure, the child's physical parameters (heart rate, respiratory rate, oxygen saturation) and anxiety will be measured and recorded. Then, the child will be shown distraction cards and inhalation therapy will be started simultaneously. Playing with the distraction cards will continue for 10 minutes until the end of the inhalation therapy. Then, the use of the toys will be stopped and the child's physiological parameters and anxiety will be recorded after 1 minute. The video recording will be ended. For participants who want to participate in the study but do not consent to being video recorded, the evaluations will be made by a nurse independent of the study.
  Arms: group of distraction cards
Other: inhalation therapy — After the consent is received, the video recording will be started. 1 minute before the procedure, the child's physical parameters (heart rate, respiratory rate, oxygen saturation) and anxiety will be measured and recorded. Then, inhalation therapy will be started with routine service application. The child will receive inhalation therapy for 10 minutes. 1 minute after the procedure, physiological parameters and anxiety will be measured and recorded again. The video recording will be ended. For participants who want to participate in the study but do not approve of being video recorded, evaluations will be made by a nurse independent of the study.
  Arms: control group

SUMMARY:
In the literature, studies examining the effect of virtual reality application on physiological parameters and anxiety during inhalation therapy, which is frequently used in children, are quite limited. Therefore, this study will be conducted to determine the effect of virtual reality goggles and distraction cards on physiological parameters and anxiety in patients receiving inhalation therapy.

DETAILED DESCRIPTION:
According to the Global Sustainable Development Report, virtual reality (VR) is one of the issues that are expected to bring about major innovations in applications, and this concept was first used by Jaron Lanier towards the end of the 1980s. VR enables computer-generated three-dimensional images and animations to interact with these objects in the environment while giving the feeling of being in a real environment in people's minds with technological tools. The purpose of VR is to make the user believe that they are in the computer-generated environment as much as possible. According to the Turkish Language Association, it is defined as 'a three-dimensional environment created by giving imitations of real environments in a virtual sphere that provides 360-degree vision using artificial intelligence, where unreal environments can be experienced as real, solving complex problems, information transfer, entertainment, etc. It is used for purposes'. Virtual reality technology is used in the field of health as a method of distraction that provides various visual, auditory, tactile and olfactory stimuli and real perceptual stimuli and is applied in many processes related to care and treatment in the health sector, especially in children. Technologies used in health care services accelerate the recovery of patients and provide ease of operation to health professionals. Children encounter many acute or chronic diseases during their developmental period. Hospitalisation as a result of these diseases is complicated and stressful for children and their families and can cause fear, anxiety and anxiety in children. Medical procedures encountered during hospitalisation are the main source of fear for children. They may experience anger, helplessness and anxiety due to reasons such as unfamiliar environment, change in the routine of the child, different sound, light, tools and equipment, unfamiliar people, painful painful procedures, being away from family and friends, loss of control, activity limitation, communication difficulties, presence of other children crying. The use of technology in preparation for or during medical procedures is an effective method in providing anxiety and comfort. Virtual reality is used in injection applications, intravenous interventions, burn dressings and postoperative pain experiences and physiological parameters in children and adolescents. Kurban and Şener investigated the effect of virtual reality goggles applied during vaccination on pain and anxiety in children aged 6-12 years and reported that the VR group had significantly lower pain and anxiety scores. In a systematic review conducted by Nacaroğlu et al. to examine the effect of virtual reality applications on pain and anxiety perception during invasive and painful procedures in school-age children in Turkey, it was reported that VR application positively affected pain and anxiety. In the study conducted by Okay and Okay in 2024 to examine the effect of virtual reality goggles on physiological parameters during inhalation therapy in children aged 2-5 years, it was observed that children watching videos with virtual reality goggles decreased the number of respirations and heart rate per minute, increased oxygen saturation values, decreased crying time and increased treatment efficacy. At the same time, although each child has different interests, it was observed that children experienced less fear and anxiety in studies where calming ocean videos were watched. Respiratory system diseases are frequently seen in childhood and constitute a significant portion of hospital admissions. Respiratory system diseases are an important cause of mortality and morbidity all over the world, a serious public health problem in developed and developing countries, and constitute 8.2% of all disabilities. According to WHO, respiratory tract infections are the most common cause of mortality in children under five years of age and are responsible for 19% of child deaths. According to the data of Turkish Statistical Institute (TurkStat), upper respiratory tract infections (URTI) are the most common disease in the 0-14 age range in our country. Inhalation therapy, which is one of the important methods in the management of respiratory system diseases, is frequently used in paediatric patients to relieve bronchospasm and to relieve the airway by delivering drug particles to the extreme lobes of the lungs. Inhalation therapy is frequently preferred because of its rapid effect, the absence of the need for an intravenous catheter and thus the absence of injection-related pain, the direct effect of the drug on the desired area (lungs), the low side effects on other systems, and the fact that it can be used at any age. Although inhalation treatment with mask is an easy intervention, it is an application that causes fear and anxiety in children. Success in treatment is ensured by the compliance of the child and the family. Children generally do not accept mask treatment and show crying and refusal behaviour. Since the crying of the child during the treatment will reduce intrapulmonary storage, the amount of drug reaching the lungs will decrease and may adversely affect the treatment. At the same time, respiratory distress experienced by children causes anxiety, dyspnoea and increase in respiratory rate. For these reasons, children receiving inhalation therapy should be calm. In order to provide effective inhalation therapy, it is recommended to use evidence-based distraction methods. There are many methods used to divert attention. Some of these are; watching cartoons, hypnotherapy, playing with toys, using virtual reality goggles, music therapy, play therapy, using kaleidoscope and using distraction cards. The method used to divert the attention of paediatric patients should affect both visual and auditory senses and at the same time be appropriate for the development of the child. The aim of the paediatric nurse is to protect and improve the mental, physical, social and spiritual health of the child and to provide holistic care for treatment in the presence of disease. In the literature, studies examining the effect of virtual reality application on physiological parameters and anxiety during inhalation therapy, which is frequently used in children, are quite limited. Therefore, this study will be conducted to determine the effect of virtual reality goggles and distraction cards on physiological parameters and anxiety in patients receiving inhalation therapy.

ELIGIBILITY:
Inclusion Criteria:

* The child is receiving inhalation (salbutamol) treatment in the pediatric intensive care unit.
* The child must be between 6-12 years old
* The child must not have any vision or hearing problems.
* Being conscious and being able to communicate verbally
* After being informed, the child and parent agree to participate in the study in writing and verbally
* No genetic, congenital, chronic or metabolic disease
* The child has no signs of respiratory failure

Exclusion Criteria:

* The child's clinical treatment is due to a history of surgery,
* The child is taking a sedative medication,
* The child has a fever over 37°C,
* The child has applied with a severe asthma attack,
* The child's saturation value is below 92% at the time of application.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Children's Emotional Manifestation Scale-CEMS | 1 minute before and 10 minutes after the start of the procedure and for approximately 1 year
  This scale was developed by William Li and Lopez in 2003 to assess the anxiety level in children aged 7-12. The Turkish validity and reliability of the scale was conducted by Yanık et al. in 2019, after receiving the approval and opinion of William Li and Lopez regarding the suitability of assessing anxiety in children aged 3-6. The scale has 5 different categories and 25 items and is used to assess the anxiety level of children aged 3-12 during medical interventions. The child's facial expressions are assessed in the facial expression category. Tears are assessed in the vocalization category. Evaluation is made according to the child's body language in the movement category. The child's verbal/nonverbal communication is assessed in the interaction category. The child's active/passive participation is assessed in the cooperation category. Each category is between 1-5 points and a total score of 5-25 points is obtained.

IPD SHARING:
Plan to Share IPD: No
I can share it when necessary, I'm not thinking about it right now.